CLINICAL TRIAL: NCT03100409
Title: Effect of a Low Residue Diet in Comparison to the Dietary Recommendations From the INCan: A Randomized Clinical Trial to Assess Malnutrition, Gastrointestinal Toxicity and Quality of Life of Advanced Cervical Cancer Patients (IB2-IVA)
Brief Title: Effect of a Low Residue Diet in Comparison to the Dietetic Recommendations From the INCan in Cervical Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was closed prematurely because the interim analysis found that subjects in the experimental group had less gastrointestinal toxicity.
Sponsor: National Institute of Cancerología (Other Government)
Collaborators: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Dr. Lucely Cetina Pérez, MD, MSc., National Institute of Cancerología
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: CEI/1125/17; INCAN (Other: Instituto Nacional de Cancerología)
Record Dates: First submitted 2017-03-24; First posted 2017-04-04 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Uterine Cervical Neoplasm; Dietary Modification; Radiation Toxicity; Gastrointestinal Complication
Keywords: Cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Radiation Injuries | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary modification (Experimental): Personalized dietary intervention, low residue diet
  Interventions: Other: Dietary modification
- Control (No Intervention): Dietary recommendations currently used in the INCan

INTERVENTIONS:
Other: Dietary modification — Dietary intervention will consist on a low residue diet: 20% kcal from fat, 5g lactose/day, 20g fiber/day (5g from insoluble fiber).
  Dietary intervention will be adapted to the patient's individual requirements, according to the presence of comorbidities or renal deterioration.
  1. No comorbidities. Energy: 20-30 kcal/kg of body weight/day. Protein: 1.3 g/kg of body weight/day.
  2. Comorbidities (diabetes, hypertension), or geriatric patient. Energy: 25-30 kcal/kg of body weight/day. Protein: 1.5 g/kg of body weight/day.
  3. Renal deterioration. Energy: 30-35 kcal/kg of body weight/day. Protein: 1 g/kg of body weight/day. Sodium: 2000-2300 mg/day. Potassium: 1900-2730 mg/day. Phosphorus: 800-1000 mg/day.
  Arms: Dietary modification

SUMMARY:
In Mexico, cervical cancer (CC) ranks second in incidence and mortality among women. The National Institute of Cancer in Mexico (lNCan) receives annually about 500 patients with CC, 80% of which are diagnosed with locally advanced disease. The standard treatment for locally advanced disease consists in concomitant chemo-radiotherapy based on cisplatin (QT-RT), followed by brachytherapy, with an absolute benefit of 10%. Adverse effects include gastrointestinal toxicity, which is the most important factor limiting the dosage of pelvic radiation. Cancer treatment, in any modality, induces malnutrition, more so when combined treatments are administered. Radiation induced gastrointestinal toxicity is caused by different factors, among which are malabsorption of bile, fat and carbohydrates, decrease in brush border enzymes, diverticular disease, proctitis, and psychological factors. International guidelines for cancer patients recommend nutritional assessment in these patients before they start treatment, so nutritional risk can be detected and the patient may get started on dietary intervention to prevent malnutrition. Several authors have studied the dietary management that may help reduce the gastrointestinal effects in cancer patients receiving pelvic radiotherapy. To reduce diarrhea and prevent malnutrition the recommended dietary approach is a low residue diet consisting on 20-25% kcal from fat, 5g of lactose and 20g of fiber. Currently the INCan does not follow the nutrition care process for cervical cancer patients; written recommendations are given to the patients with a list of foods allowed or not allowed, with no further nutritional assessment or intervention. From previous studies, the investigators have demonstrated that the current recommendations do not help the patients maintain their nutritional status, during their treatment most patients become malnourished (81%, p<0.01). Therefore, the aim of this clinical trial is to evaluate a diet low in residue in CC patients, considering the necessary modifications for each patient if morbidities are present, in comparison with the current dietary recommendations used in the INCan.

DETAILED DESCRIPTION:
In Mexico, cervical cancer (CC) is the second most frequent cause of death among women, with a mortality rate of 4000 women/year. Among the patients attended by the INCan, 80% are diagnosed with locally advanced CC and 30% of these present comorbidities. Hypertension may be present in 20% of patients, obesity in 18% and diabetes in 6.8%. These comorbidities affect the efficacy of treatment, increase the risk of malnutrition, of adverse events, hospitalization, increase hospital stay and worsen the quality of life, and even increase the risk of death. Furthermore, 10 to 20% of patients present kidney deterioration. The main reason for kidney disease is ureteral obstruction. The glomerular filtration rate deteriorates with age and many patients have comorbid medical illnesses that further compromise the kidneys. The standard treatment for CC is concomitant chemo-radiotherapy using cisplatin as a radiosensitizer, and brachytherapy at the end of treatment. Studies developed in the INCan described the acute toxicity symptoms in CC patients using this treatment: nausea, vomiting, diarrhea, cystitis, radioepithelitis, leucopenia, neutropenia, thrombocytopenia. Pelvic radiotherapy causes gastrointestinal toxicity, which is the most important limiting factor for the patients to complete their treatment. Cancer treatment, along with the tumor itself and other factors, causes malnutrition, and this confers a bad prognosis for the patient's response to treatment and survival. There is a nutritional risk in these patients at the moment of diagnosis, because of the metabolic alterations caused by the tumor, and the treatment-induced side effects. International guidelines for cancer patients recommend nutritional assessment in these patients before they start treatment, so nutritional risk can be detected and the patient may get started on dietary intervention to prevent malnutrition. Several authors have studied the dietary management that may help reduce the gastrointestinal effects in cancer patients receiving pelvic radiotherapy. To reduce diarrhea and prevent malnutrition the recommended dietary approach is a low residue diet consisting on 20-25% fat, 5g of lactose and 20g of fiber. Currently the INCan does not follow the nutrition care process for cervical cancer patients; written recommendations are given to the patients with a list of foods allowed or not allowed, with no further nutritional assessment or intervention. The investigators described the nutritional status of CC patients undergoing concomitant chemo-radiotherapy. It was observed that by the end of cancer treatment, a period of 9 weeks, 81.8% of patients became malnourished; 96% of patients lost weight, 78% of which had severe weight loss.

The aim of this clinical trial is to evaluate a diet low in residue in CC patients, considering the necessary modifications for each patient if morbidities are present, in comparison with the current dietary recommendations used in the INCan. A thorough nutritional evaluation including anthropometric data, dietary data, gastrointestinal toxicity and quality of life evaluations, will be performed.

Particular objectives are the following:

1. Identify the nutritional status of CC patients before, during and after treatment with chemo-radiotherapy, in intervention and control groups.
2. Determine the association of malnutrition and gastrointestinal toxicity during and after treatment, in intervention and control groups.
3. Evaluate the quality of life of patients before, during and after treatment, in both groups.
4. Establish the association of nutritional status and response to treatment, in both groups.

The aim is based on the following hypothesis: Patients receiving the personalized nutritional intervention with the low residue diet will maintain a better nutritional status during treatment, reflected in fewer malnourished patients, compared to the control group.

Methods.

Study design. Randomized clinical trial, open, factorial 3X2. To evaluate the efficacy of a low residue diet on the nutritional status, gastrointestinal toxicity and quality of life of CC patients referring to the National Institute of Cancer in Mexico (INCan). 320 patients will be included, with cervical malignant tumors of epithelial origin in the neck of the uterus, candidates for chemo-radiotherapy.

Dietary intervention will consist on a low residue diet: 20% kcal from fat, 5g lactose/day, 20g fiber/day (5g from insoluble fiber).

Dietary intervention will be adapted to the patient's individual requirements, according to the presence of comorbidities or renal deterioration.

1. No comorbidities. Energy: 20-30 kcal/kg of body weight/day. Protein: 1.3 g/kg of body weight/day.
2. Comorbidities (diabetes, hypertension), or geriatric patient. Energy: 25-30 kcal/kg of body weight/day. Protein: 1.5 g/kg of body weight/day.
3. Renal deterioration.

Energy: 30-35 kcal/kg of body weight/day.

Protein: 1 g/kg of body weight/day.

Sodium: 2000-2300 mg/day

Potassium: 1900-2730 mg/day

Phosphorus: 800-1000 mg/day

Control group will receive the standard written recommendations from the INCan, which enlist allowed foods and not allowed foods.

Sample size.

A sample space of 320 patients will be included if prior consent is acquired and if they meet the inclusion criteria. This clinical trial contemplates 3 strata with 2 levels.

Statistical analysis.

A univariate analysis will be performed to describe the study population. Descriptive statistics will be used to obtain measures of central tendency and dispersion, as well as frequency of distribution for qualitative variables. Percentage change of nutritional status will be calculated using the Friedman test. Chi square test will be used to compare basal vs final assessment, and chi square test will be used to compare among study groups. All confidence intervals will be constructed with a confidence of 95% (α=0.05). The interpretation of the study results will be responsibility of researchers. Data processing and analysis will be performed with the SPSS package (version 19.0®) for Microsoft.

Efficacy analysis.

Efficacy will be evaluated in patients that qualify to be included in the protocol analysis. To evaluate efficacy, nutritional diagnosis through the clinical course will be analyzed in both, intervention and control, groups. Also, toxicity and quality of life responses will be obtained.

Procedures.

Treatment. Anticancer treatment will consist of Cisplatin as a radiosensitizer, at a dosage of 40 mg/m2/week for 6 weeks. For patients with renal deterioration Gemcitabine will be used instead of Cisplatin, at a dosage of 300 mg/m2/week for 6 weeks. Concomitantly, external pelvic radiotherapy will be applied at a total dosage of 50.4 Gy divided by 28 fractions, 1.8 Gy/day/5 days a week, for 6 weeks. After completing concomitant chemo-radiotherapy, intracavitary brachytherapy will be administered at low dosage (30 Gy of Cesium 137) or high dosage (Iridium). Before initiating chemo-radiotherapy, a complete evaluation will be applied as mentioned.

Once eligibility criteria are verified, patients will be randomly assigned to intervention group or control group.

Visits during the study. After signing the informed consent, the patient will be informed when she will begin participating in the study (screening visit). If the patient complies with the inclusion criteria, a total of 5 visits will be scheduled: (1) at week -2, 2 weeks before treatment; (2) at week 0, on initiation of treatment; (3) at week 3, on the 3rd cycle of chemotherapy; (4) at week 9, by the end of brachytherapy; and (5) at week 21, 3 months after treatment completion.

Monitoring.

A thorough evaluation on each visit will be performed using the following tools:

* Patient generated subjective global assessment.
* Anthropometric data: weight, height, waist circumference, hip circumference, arm circumference.
* Body mass index.
* Waist to hip ratio.
* Body composition (bioelectrical impedance).
* % weight loss.
* Hand dynamometry.
* Dietary data: 24 hour recall and frequency of food intake questionnaires.
* % recommended energy intake.
* Biochemical markers: serum albumin, number of lymphocytes.
* Gastrointestinal toxicity using the CTCAE v4.03.
* Quality of life using the QLQ-C30 and CxC24.

Sample collection. No tissue or additional blood samples will be obtained, other than the blood samples used as part of the routine clinical laboratory tests.

Informed consent acquisition. On the screening visit, the written consent will be read and explained to the patient, clarifying the risks and benefits involved in the study. Two witnesses, independent from the study, will be present. The patient will have the choice to not participate or withdraw from the study at any time, her decision will not affect the quality of care and treatment that the attending physician will provide. The researcher will be governed by the ethical principles established in the Helsinki Accord. The physician will adequately respond all the matters of interest to the patient.

Ethical considerations.

The Research Committee and the Ethics Committee of the National Institute of Cancer in Mexico has approved the protocol and the informed consent document.

Patients participating in this study will be informed, through the informed consent, of all the details concerning this trial. The patients who agree to participate in the trial will express their willingness by signing the informed consent document, being clarified that they can leave the trial at any time, if they wish to do so.

Regulatory considerations.

This study abides by the ethical principles established by the international community, in accordance to the Good Clinical Practices, the Nüremberg Code, the Helsinki Accord, the Statement of Compliance with International Conference on Harmonization Guidelines for Good Clinical Practice, and the Regulations of the General Law of Health in the matter of research for health.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age and older.
* Ability to understand the study and be able to sign the informed consent.
* Functional stage ECOG 0 - 2.
* Negative pregnancy test, null reproductive potential, or currently using an contraceptive method.
* Willing and able to attend the programmed visits.
* Diagnosed with cervical malignant tumors of epithelial origin in the neck of the uterus, clinical stages IB2-IVA.
* Candidates to receive concomitant Chemo-Radiotherapy, followed by Brachytherapy.
* In case of presence of diabetes mellitus and/or hypertension, without retinopathy or albuminuria <300 mg/dl.
* In case of renal deterioration, a creatinine clearance >20 ml/min.
* Hemoglobin >10 g/l.
* Leucocytes > 4000/mm3.
* Platelets >100000/mm3.

Exclusion Criteria:

* Under a different nutritional treatment using a nutritional supplement.
* Carrying other uncontrolled diseases, including cardiovascular insufficiency, arrhythmia, psychiatric illnesses.
* Concomitant treatment with another experimental drug.
* Active TB.
* Infected with HIV.
* History of LES and other rheumatologic diseases that involve renal deterioration.
* Presence of vesicular-vaginal fistulae at moment of diagnosis.
* Previous malignancy.

Study Discontinuation Criteria:

* Loss of follow up for 21 days.
* Evidence of disease progression.
* At the request of patient.
* By unacceptable toxicity.
* Pregnancy.

Criteria must be followed punctually. If a patient were inappropriately included, she must be discontinued from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Gastrointestinal toxicity symptoms grading scale using the Common Toxicity Criteria for Adverse Events (CTCAE v4) | Baseline, 3 weeks after treatment initiation, 12 weeks after treatment initiation and 6 months after treatment initiation .
  Evaluation of the gastrointestinal symptoms according to the Common Toxicity Criteria for Adverse Events (CTCAE v4).
  A grading scale is provided for each adverse event (AE) term. Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living.
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Changes in nutritional status | Baseline, 3 weeks after treatment initiation, 12 weeks after treatment initiation and 6 months after treatment initiation .
  Evaluation the change of the nutritional status by the Patient Generated Subjective Global Assessment.
  The Patient Generated Subjective Global Assessment is a questionnaire that comprises 7 sections: weight, intake, symptoms, functional capacity, disease and its relationship to nutritional requirements, metabolic demand and physical evaluation. Based on the previous results the interviewer will define which of the following three groups the individual surveyed belongs to:
  A: well nourished. B: moderately or suspiciously undernourished. C: severely malnourished.
Changes in food intake | Baseline, 3 weeks after treatment initiation, 12 weeks after treatment initiation and 6 months after treatment initiation .
  Change in food intake assessed by 24-hour reminder This method consists of questioning the subject to find out everything he or she ingested the day before. It includes three lists of foods to help the interviewee remember, the first is a quick list that contains drinks and foods, the second list contains foods that are commonly forgotten and the interview closes with a detailed description of everything that was consumed

SECONDARY OUTCOMES:
Changes in body weight | Baseline, 3 weeks after treatment initiation, 12 weeks after treatment initiation and 6 months after treatment initiation .
  Evaluation the changes of the body weight (kilograms) The measurement will be done on a hospital scale SECA brand.
Changes in body composition (phase angle) | Baseline, 3 weeks after treatment initiation, 12 weeks after treatment initiation and 6 months after treatment initiation .
  Evaluation the changes of the phase angle (grades) by the bioelectrical impedance Biolelectrical impedances will be evaluated by body composition analyzer Quantun IV The phase angle is a nutritional indicator which evaluates the distribution of intracellular and extracellular fluid, therefore, it has been described as an indicator of the quality of the cell membrane
Changes in handgrip strength measures | Baseline, 3 weeks after treatment initiation, 12 weeks after treatment initiation and 6 months after treatment initiation .
  Evaluation the change of the handgrip strength (kilograms)
  Handgript strength will be evaluated by a dinamometer Takei Hand strength is a simple measure, it has been used to estimate total muscle strength and has been described as a marker of nutritional status, in addition, it is related to mortality and morbidity (56).
  The instrument for measuring hand force is the dynamometer, and the cut-off points for making a diagnosis of sarcopenia in women is a result ﹤de 20 kg, while in men it is ﹤de 30 kg
Change in quality of life summary score using the the quality of life questionnaire specifically developed for cancer patients (European Organization for Research and Treatment of Cancer Core 30 (EORTC QLQ-C30 v3)) | Baseline, 3 weeks after treatment initiation, 12 weeks after treatment initiation and 6 months after treatment initiation .
  Quality of life questionnaire developed and validated for cancer patients ((European Organization for Research and Treatment of Cancer Core 30 (EORTC QLQ-C30 v3)) will be applied, and the change in summary score will be evaluated.
  The EORTC QLQ-C30 questionnaire evaluates the quality of life in oncological population, is composed of both multi-item and single-item measures. It has 30 items, including nine scales: five functional scales (physical, role, emotional, cognitive and social functioning), three symptom scales (fatigue, pain and nausea / vomiting) and one global health status/QoL scale. Six single items are also included (Dyspnea, Insomnia, Appetite loss, Constipation, Diarrhea and Financial difficulties). A high score for all functional and global health/QoL scales represents a high/healthy level of functioning/high QoL, whereas a high score for a symptom scale/item represents a high level of symptoms/problems.
Change in quality of life for cervical cancer patients: (European Organization for Research and Treatment of Cancer Cervical cancer module- EORTC QLQ-CX 24) | Baseline, 3 weeks after treatment initiation, 12 weeks after treatment initiation and 6 months after treatment initiation .
  Change in quality of life summary score and subescales using The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Cervical Cancer Module (EORTC QLQ-CX24). The EORTC QLQ-CX24 is the supplementary module of the QLQ-C30 aimed to evaluate quality of life of cervical cancer patients.
  The EORTC QLQ-CX24 is the supplementary module of the QLQ-C30 aimed to evaluate quality of life of cervical cancer patients. It consists of 24 items divided in three multi-item scales to assess symptoms experience (gastrointestinal and genitourinary), body image and sexual/vaginal functioning, and six single items to assess lymphedema, peripheral neuropathy, menopausal symptoms, sexual worry, sexual activity and sexual enjoyment. The last five questions are answered only by patients with an active sex life. Higher scores are equivalent to worse or more symptoms, except for items 49 and 54 (higher score indicates better quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Lucely C Cetina, MD, MSc, Principal Investigator — National Institute of Cancerología
Locations (1):
- National Cancer Institute of Mexico, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Argiles JM. Cancer-associated malnutrition. Eur J Oncol Nurs. 2005;9 Suppl 2:S39-50. doi: 10.1016/j.ejon.2005.09.006. PMID 16437757
- [Background] Arrieta O, Michel Ortega RM, Villanueva-Rodriguez G, Serna-Thome MG, Flores-Estrada D, Diaz-Romero C, Rodriguez CM, Martinez L, Sanchez-Lara K. Association of nutritional status and serum albumin levels with development of toxicity in patients with advanced non-small cell lung cancer treated with paclitaxel-cisplatin chemotherapy: a prospective study. BMC Cancer. 2010 Feb 21;10:50. doi: 10.1186/1471-2407-10-50. PMID 20170547
- [Background] Bantle JP, Wylie-Rosett J, Albright AL, Apovian CM, Clark NG, Franz MJ, Hoogwerf BJ, Lichtenstein AH, Mayer-Davis E, Mooradian AD, Wheeler ML. Nutrition recommendations and interventions for diabetes--2006: a position statement of the American Diabetes Association. Diabetes Care. 2006 Sep;29(9):2140-57. doi: 10.2337/dc06-9914. No abstract available. PMID 16936169
- [Background] Beale RJ, Bryg DJ, Bihari DJ. Immunonutrition in the critically ill: a systematic review of clinical outcome. Crit Care Med. 1999 Dec;27(12):2799-805. doi: 10.1097/00003246-199912000-00032. PMID 10628629
- [Background] Bye A, Kaasa S, Ose T, Sundfor K, Trope C. The influence of low fat, low lactose diet on diarrhoea during pelvic radiotherapy. Clin Nutr. 1992 Jun;11(3):147-53. doi: 10.1016/0261-5614(92)90075-2. PMID 16839990
- [Background] Calder PC, Kew S. The immune system: a target for functional foods? Br J Nutr. 2002 Nov;88 Suppl 2:S165-77. doi: 10.1079/BJN2002682. PMID 12495459
- [Background] Capra S, Ferguson M, Ried K. Cancer: impact of nutrition intervention outcome--nutrition issues for patients. Nutrition. 2001 Sep;17(9):769-72. doi: 10.1016/s0899-9007(01)00632-3. PMID 11527676
- [Background] Chandra RK. Nutrition and the immune system: an introduction. Am J Clin Nutr. 1997 Aug;66(2):460S-463S. doi: 10.1093/ajcn/66.2.460S. PMID 9250133
- [Background] Rock CL, Moskowitz A, Huizar B, Saenz CC, Clark JT, Daly TL, Chin H, Behling C, Ruffin MT 4th. High vegetable and fruit diet intervention in premenopausal women with cervical intraepithelial neoplasia. J Am Diet Assoc. 2001 Oct;101(10):1167-74. doi: 10.1016/S0002-8223(01)00286-3. PMID 11678487
- [Background] Coia LR, Myerson RJ, Tepper JE. Late effects of radiation therapy on the gastrointestinal tract. Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1213-36. doi: 10.1016/0360-3016(94)00419-L. PMID 7713784
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Pia de la Maza M, Agudelo GM, Yudin T, Gattas V, Barrera G, Bunout D, Hirsch S. Long-term nutritional and digestive consequences of pelvic radiation. J Am Coll Nutr. 2004 Apr;23(2):102-7. doi: 10.1080/07315724.2004.10719349. PMID 15047675
- [Background] Pia de la Maza M, Gotteland M, Ramirez C, Araya M, Yudin T, Bunout D, Hirsch S. Acute nutritional and intestinal changes after pelvic radiation. J Am Coll Nutr. 2001 Dec;20(6):637-42. doi: 10.1080/07315724.2001.10719161. PMID 11771680
- [Background] Shin DW, Nam JH, Kwon YC, Park SY, Bae DS, Park CT, Cho CH, Lee JM, Park SM, Yun YH. Comorbidity in disease-free survivors of cervical cancer compared with the general female population. Oncology. 2008;74(3-4):207-15. doi: 10.1159/000151368. Epub 2008 Aug 20. PMID 18714169
- [Background] Duenas-Gonzalez A, Lopez-Graniel C, Gonzalez-Enciso A, Cetina L, Rivera L, Mariscal I, Montalvo G, Gomez E, de la Garza J, Chanona G, Mohar A. A phase II study of multimodality treatment for locally advanced cervical cancer: neoadjuvant carboplatin and paclitaxel followed by radical hysterectomy and adjuvant cisplatin chemoradiation. Ann Oncol. 2003 Aug;14(8):1278-84. doi: 10.1093/annonc/mdg333. PMID 12881393
- [Background] Duenas-Gonzalez A, Cetina L, Sanchez B, Gomez E, Rivera L, Hinojosa J, Lopez-Graniel C, Gonzalez-Enciso A, de la Garza J. A phase I study of carboplatin concurrent with radiation in FIGO stage IIIB cervix uteri carcinoma. Int J Radiat Oncol Biol Phys. 2003 Aug 1;56(5):1361-5. doi: 10.1016/s0360-3016(03)00347-x. PMID 12873681
- [Background] Arends J, Bodoky G, Bozzetti F, Fearon K, Muscaritoli M, Selga G, van Bokhorst-de van der Schueren MA, von Meyenfeldt M; DGEM (German Society for Nutritional Medicine); Zurcher G, Fietkau R, Aulbert E, Frick B, Holm M, Kneba M, Mestrom HJ, Zander A; ESPEN (European Society for Parenteral and Enteral Nutrition). ESPEN Guidelines on Enteral Nutrition: Non-surgical oncology. Clin Nutr. 2006 Apr;25(2):245-59. doi: 10.1016/j.clnu.2006.01.020. Epub 2006 May 12. PMID 16697500
- [Background] Fearon KC, Moses AG. Cancer cachexia. Int J Cardiol. 2002 Sep;85(1):73-81. doi: 10.1016/s0167-5273(02)00235-8. PMID 12163211
- [Background] Gomez-Candela C, Luengo LM, Cos AI, Martinez-Roque V, Iglesias C, Zamora P, Gonzalez-Baron R. [Subjective global assessment in neoplastic patients]. Nutr Hosp. 2003 Nov-Dec;18(6):353-7. Spanish. PMID 14682183
- [Background] Garcia-Luna PP, Parejo Campos J, Pereira Cunill JL. [Causes and impact of hyponutrition and cachexia in the oncologic patient]. Nutr Hosp. 2006 May;21 Suppl 3:10-6. Spanish. PMID 16768026
- [Background] Gonzalez-Pinto I, Gonzalez EM. Optimising the treatment of upper gastrointestinal fistulae. Gut. 2001 Dec;49 Suppl 4(Suppl 4):iv22-31. doi: 10.1136/gut.49.suppl_4.iv21. PMID 11878791
- [Background] Henson CC, Burden S, Davidson SE, Lal S. Nutritional interventions for reducing gastrointestinal toxicity in adults undergoing radical pelvic radiotherapy. Cochrane Database Syst Rev. 2013 Nov 26;2013(11):CD009896. doi: 10.1002/14651858.CD009896.pub2. PMID 24282062
- [Background] Hernandez-Avila M, Romieu I, Parra S, Hernandez-Avila J, Madrigal H, Willett W. Validity and reproducibility of a food frequency questionnaire to assess dietary intake of women living in Mexico City. Salud Publica Mex. 1998 Mar-Apr;40(2):133-40. doi: 10.1590/s0036-36341998000200005. PMID 9617194
- [Background] Inagaki J, Rodriguez V, Bodey GP. Proceedings: Causes of death in cancer patients. Cancer. 1974 Feb;33(2):568-73. doi: 10.1002/1097-0142(197402)33:23.0.co;2-2. No abstract available. PMID 4591273
- [Background] Isenring EA, Capra S, Bauer JD. Nutrition intervention is beneficial in oncology outpatients receiving radiotherapy to the gastrointestinal or head and neck area. Br J Cancer. 2004 Aug 2;91(3):447-52. doi: 10.1038/sj.bjc.6601962. PMID 15226773
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Kizer NT, Thaker PH, Gao F, Zighelboim I, Powell MA, Rader JS, Mutch DG, Grigsby PW. The effects of body mass index on complications and survival outcomes in patients with cervical carcinoma undergoing curative chemoradiation therapy. Cancer. 2011 Mar 1;117(5):948-56. doi: 10.1002/cncr.25544. Epub 2010 Oct 13. PMID 20945318
- [Background] Krauss RM, Eckel RH, Howard B, Appel LJ, Daniels SR, Deckelbaum RJ, Erdman JW Jr, Kris-Etherton P, Goldberg IJ, Kotchen TA, Lichtenstein AH, Mitch WE, Mullis R, Robinson K, Wylie-Rosett J, St Jeor S, Suttie J, Tribble DL, Bazzarre TL. AHA Dietary Guidelines: revision 2000: A statement for healthcare professionals from the Nutrition Committee of the American Heart Association. Circulation. 2000 Oct 31;102(18):2284-99. doi: 10.1161/01.cir.102.18.2284. No abstract available. PMID 11056107
- [Background] Kuenstner S, Langelotz C, Budach V, Possinger K, Krause B, Sezer O. The comparability of quality of life scores. a multitrait multimethod analysis of the EORTC QLQ-C30, SF-36 and FLIC questionnaires. Eur J Cancer. 2002 Feb;38(3):339-48. doi: 10.1016/s0959-8049(01)00369-0. PMID 11818198
- [Background] Le T, Hopkins L, Kee Fung MF. Quality of life assessment during adjuvant and salvage chemotherapy for advance stage epithelial ovarian cancer. Gynecol Oncol. 2005 Jul;98(1):39-44. doi: 10.1016/j.ygyno.2005.03.040. PMID 15907986
- [Background] Levine MN, Ganz PA. Beyond the development of quality-of-life instruments: where do we go from here? J Clin Oncol. 2002 May 1;20(9):2215-6. doi: 10.1200/JCO.2002.20.9.2215. No abstract available. PMID 11980989
- [Background] Mohar A, Frias-Mendivil M. Epidemiology of cervical cancer. Cancer Invest. 2000;18(6):584-90. doi: 10.3109/07357900009012198. No abstract available. PMID 10923107
- [Background] Movsas B. Quality of life in oncology trials: a clinical guide. Semin Radiat Oncol. 2003 Jul;13(3):235-47. doi: 10.1016/S1053-4296(03)00029-8. PMID 12903013
- [Background] Murphy J, Stacey D, Crook J, Thompson B, Panetta D. Testing control of radiation-induced diarrhea with a psyllium bulking agent: a pilot study. Can Oncol Nurs J. 2000 Summer;10(3):96-100. doi: 10.5737/1181912x10396100. PMID 11894282
- [Background] Obarzanek E, Sacks FM, Vollmer WM, Bray GA, Miller ER 3rd, Lin PH, Karanja NM, Most-Windhauser MM, Moore TJ, Swain JF, Bales CW, Proschan MA; DASH Research Group. Effects on blood lipids of a blood pressure-lowering diet: the Dietary Approaches to Stop Hypertension (DASH) Trial. Am J Clin Nutr. 2001 Jul;74(1):80-9. doi: 10.1093/ajcn/74.1.80. PMID 11451721
- [Background] Obermair A, Hagenauer S, Tamandl D, Clayton RD, Nicklin JL, Perrin LC, Ward BG, Crandon AJ. Safety and efficacy of low anterior en bloc resection as part of cytoreductive surgery for patients with ovarian cancer. Gynecol Oncol. 2001 Oct;83(1):115-20. doi: 10.1006/gyno.2001.6353. PMID 11585422
- [Background] Paddon-Jones D, Short KR, Campbell WW, Volpi E, Wolfe RR. Role of dietary protein in the sarcopenia of aging. Am J Clin Nutr. 2008 May;87(5):1562S-1566S. doi: 10.1093/ajcn/87.5.1562S. PMID 18469288
- [Background] Pearcey R, Brundage M, Drouin P, Jeffrey J, Johnston D, Lukka H, MacLean G, Souhami L, Stuart G, Tu D. Phase III trial comparing radical radiotherapy with and without cisplatin chemotherapy in patients with advanced squamous cell cancer of the cervix. J Clin Oncol. 2002 Feb 15;20(4):966-72. doi: 10.1200/JCO.2002.20.4.966. PMID 11844818
- [Background] Pettersson A, Nygren P, Persson C, Berglund A, Turesson I, Johansson B. Effects of a dietary intervention on gastrointestinal symptoms after prostate cancer radiotherapy: long-term results from a randomized controlled trial. Radiother Oncol. 2014 Nov;113(2):240-7. doi: 10.1016/j.radonc.2014.11.025. Epub 2014 Nov 29. PMID 25467005
- [Background] Ravasco P, Monteiro-Grillo I, Vidal PM, Camilo ME. Cancer: disease and nutrition are key determinants of patients' quality of life. Support Care Cancer. 2004 Apr;12(4):246-52. doi: 10.1007/s00520-003-0568-z. Epub 2004 Mar 3. PMID 14997369
- [Background] Roberts KB, Urdaneta N, Vera R, Vera A, Gutierrez E, Aguilar Y, Ott S, Medina I, Sempere P, Rockwell S, Sartorelli AC, Fischer DB, Fischer JJ. Interim results of a randomized trial of mitomycin C as an adjunct to radical radiotherapy in the treatment of locally advanced squamous-cell carcinoma of the cervix. Int J Cancer. 2000 Aug 20;90(4):206-23. doi: 10.1002/1097-0215(20000820)90:43.0.co;2-o. PMID 10993961
- [Background] Roila F, Cortesi E. Quality of life as a primary end point in oncology. Ann Oncol. 2001;12 Suppl 3:S3-6. doi: 10.1093/annonc/12.suppl_3.s3. PMID 11804381
- [Background] Rose PG, Ali S, Watkins E, Thigpen JT, Deppe G, Clarke-Pearson DL, Insalaco S; Gynecologic Oncology Group. Long-term follow-up of a randomized trial comparing concurrent single agent cisplatin, cisplatin-based combination chemotherapy, or hydroxyurea during pelvic irradiation for locally advanced cervical cancer: a Gynecologic Oncology Group Study. J Clin Oncol. 2007 Jul 1;25(19):2804-10. doi: 10.1200/JCO.2006.09.4532. Epub 2007 May 14. PMID 17502627
- [Background] Santoso JT, Canada T, Latson B, Aaaadi K, Lucci JA 3rd, Coleman RL. Prognostic nutritional index in relation to hospital stay in women with gynecologic cancer. Obstet Gynecol. 2000 Jun;95(6 Pt 1):844-6. doi: 10.1016/s0029-7844(99)00658-4. PMID 10831978
- [Background] Santoso JT, Cannada T, O'Farrel B, Alladi K, Coleman RL. Subjective versus objective nutritional assessment study in women with gynecological cancer: a prospective cohort trial. Int J Gynecol Cancer. 2004 Mar-Apr;14(2):220-3. doi: 10.1111/j.1048-891X.2004.014203.x. PMID 15086719
- [Background] Sayer AA, Syddall H, Martin H, Patel H, Baylis D, Cooper C. The developmental origins of sarcopenia. J Nutr Health Aging. 2008 Aug-Sep;12(7):427-32. doi: 10.1007/BF02982703. No abstract available. PMID 18615224
- [Background] Segura A, Pardo J, Jara C, Zugazabeitia L, Carulla J, de Las Penas R, Garcia-Cabrera E, Luz Azuara M, Casado J, Gomez-Candela C. An epidemiological evaluation of the prevalence of malnutrition in Spanish patients with locally advanced or metastatic cancer. Clin Nutr. 2005 Oct;24(5):801-14. doi: 10.1016/j.clnu.2005.05.001. PMID 15993517
- [Background] Spirtos NM, Ballon SC. Needle catheter jejunostomy: a controlled, prospective, randomized trial in patients with gynecologic malignancy. Am J Obstet Gynecol. 1988 Jun;158(6 Pt 1):1285-90. doi: 10.1016/0002-9378(88)90358-4. PMID 3132853
- [Background] Thompson DD. Aging and sarcopenia. J Musculoskelet Neuronal Interact. 2007 Oct-Dec;7(4):344-5. No abstract available. PMID 18094505
- [Background] Tian J, Chen JS. Nutritional status and quality of life of the gastric cancer patients in Changle County of China. World J Gastroenterol. 2005 Mar 21;11(11):1582-6. doi: 10.3748/wjg.v11.i11.1582. PMID 15786531
- [Background] Van Cutsem E, Arends J. The causes and consequences of cancer-associated malnutrition. Eur J Oncol Nurs. 2005;9 Suppl 2:S51-63. doi: 10.1016/j.ejon.2005.09.007. PMID 16437758
- [Background] Wedlake LJ, McGough C, Shaw C, Klopper T, Thomas K, Lalji A, Dearnaley DP, Blake P, Tait D, Khoo VS, Andreyev HJ. Clinical trial: Efficacy of a low or modified fat diet for the prevention of gastrointestinal toxicity in patients receiving radiotherapy treatment for pelvic malignancies. J Hum Nutr Diet. 2012 Jun;25(3):247-59. doi: 10.1111/j.1365-277X.2012.01248.x. Epub 2012 Apr 20. PMID 22515941
- [Background] Whitney CW, Sause W, Bundy BN, Malfetano JH, Hannigan EV, Fowler WC Jr, Clarke-Pearson DL, Liao SY. Randomized comparison of fluorouracil plus cisplatin versus hydroxyurea as an adjunct to radiation therapy in stage IIB-IVA carcinoma of the cervix with negative para-aortic lymph nodes: a Gynecologic Oncology Group and Southwest Oncology Group study. J Clin Oncol. 1999 May;17(5):1339-48. doi: 10.1200/JCO.1999.17.5.1339. PMID 10334517
- [Background] Wong LC, Ngan HY, Cheung AN, Cheng DK, Ng TY, Choy DT. Chemoradiation and adjuvant chemotherapy in cervical cancer. J Clin Oncol. 1999 Jul;17(7):2055-60. doi: 10.1200/JCO.1999.17.7.2055. PMID 10561258
- [Background] Xue H, Sawyer MB, Wischmeyer PE, Baracos VE. Nutrition modulation of gastrointestinal toxicity related to cancer chemotherapy: from preclinical findings to clinical strategy. JPEN J Parenter Enteral Nutr. 2011 Jan;35(1):74-90. doi: 10.1177/0148607110377338. PMID 21224434
- [Result] Nagle CM, Purdie DM, Webb PM, Green A, Harvey PW, Bain CJ. Dietary influences on survival after ovarian cancer. Int J Cancer. 2003 Aug 20;106(2):264-9. doi: 10.1002/ijc.11204. PMID 12800204